CLINICAL TRIAL: NCT05304039
Title: Phenotyping and Classifying of Childhood and Adult Asthma Exacerbations: Towards Personalised Treatment. An Observational Multicentre Study.
Brief Title: Phenotyping and Classifying Asthma Exacerbations
Acronym: ExCluSieF
Status: Active, not recruiting | Type: Observational
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Erasmus Medical Center (Other); TNO (Other)
Responsible Party: Sponsor
Other Study IDs: NL79257.100.21
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Asthma Attack
Keywords: Asthma; Exacerbation; Phenotyping; Classification; Treatment
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires; Spirometry; Fractional Exhaled Nitric Oxide Testing; Electronic Nose; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Nasopharyngeal swabs Nasal lining fluid Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asthma exacerbation: Patients with an asthma exacerbation who are diagnosed with mild to severe asthma according to the GINA guidelines
  Interventions: Behavioral: Questionnaires; Device: Spirometry; Device: Fractional Exhaled Nitric Oxide (FeNO); Device: Corsano watch; Device: e-Nose; Procedure: Nasopharyngeal swabs and nasal lining fluid; Device: Sputum culture; Procedure: Blood sample

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires about asthma control and quality of life
Device: Spirometry — Spirometry monitoring at home
Device: Fractional Exhaled Nitric Oxide (FeNO) — Measuring fractional exhaled nitric oxide at home
Device: Corsano watch — Monitoring vital parameters at home
Device: e-Nose — Breathprint will be performed using e-Nose
Procedure: Nasopharyngeal swabs and nasal lining fluid — Nasopharyngeal swabs and nasal lining fluid will be performed
Device: Sputum culture — If patients produce sputum, the sputum will be analysed
Procedure: Blood sample — Blood sample for standard care and 10 ml extra will be taken

SUMMARY:
An observational study in patients between 12 and 70 years old with an acute asthma exacerbation, to determine the relation between phenotypical characteristics and the treatment response.

DETAILED DESCRIPTION:
Rationale: Asthma is a heterogeneous inflammatory respiratory disease affecting 8 - 9% of the European population. Acute asthma exacerbation (AAE) is characterized as an acute worsening of symptoms and is treated inconsistently with steroids with or without antibiotics. In order to adjust and personalise exacerbation treatment, phenotyping and classifying of asthma exacerbations would be required. Therefore, we want to classify patients with AAEs phenotypically in relation to the treatment response.

Objective: The primary objective of the study is to determine the relationship between exacerbation treatment response at day 7 and the phenotypical characteristics of asthma exacerbations. Secondary objectives are 1) developing a prediction model based on biomarkers and/or clinical data to predict the treatment response of AAEs 2) comparing the environmental, inflammatory, microbiological and lipid parameters of patients diagnosed with asthma between exacerbation phase and recovery (baseline).

Study design: A prospective cohort multicentre study. Study population: Patients aged 12 - 70 years, diagnosed with mild to severe asthma according to the Global Initiative for Asthma (GINA) guidelines. Patients will be included at the onset of a severe asthma exacerbation.

Main study parameters/endpoints: Primary endpoint is the relation of phenotypical characteristics with treatment response at day 7, defined by 1) the physician - and patient rated global evaluation of treatment effectiveness (GETE) score 2) difference in Asthma Control Questionnaire 5 (ACQ-5) (> 0.5) 3) difference in handheld spirometry values like forced expiratory volume (FEV1 ≥ 10%). Treatment response will be classified as excellent, good, moderate or poor. Secondary endpoints are 1) a prediction model for the treatment response of AAE 2) aetiology of the AAE 3) blood and local respiratory parameters; microbiota composition; lipid metabolomics and volatile compounds composition at baseline and AAE.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with asthma according to the GINA guidelines between 12 and 70 years old. If patients are doctor's diagnosed with asthma based on clinical data, the further diagnostics will be performed to confirm the asthma diagnosis after the AAE.
* Mild to severe asthma, treated according to GINA guidelines with medium - or high dose inhaled corticosteroids (with or without LABA) or treated with a low dose inhaled corticosteroids combined LABA or leukotriene - receptor antagonist.
* Asthma exacerbation, indicated for systemic corticosteroids.
* Written personal and/or parental informed consent, prior to any study procedures.
* Eligibility and willingness to present during an asthma exacerbation at the Franciscus Gasthuis hospital.
* Ability to use e - health applications.

Exclusion Criteria:

* Immunosuppressive maintenance medication (azithromycin, systemic corticosteroids maintenance therapy and other) or recently (< 6 weeks) discontinued these medications. (Desensitization therapy indicated for allergies can be included in the study)
* Maintenance medication or recently discontinued (< 6 weeks) biologicals.
* Other underlying inflammatory or auto-immune diseases, such as rheumatologic disease.
* Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site)
* Pregnancy, because of the possible altered immunological status.(31)
* Participation in an interventional study or randomised controlled trial.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 12 - 70 years, diagnosed with mild to severe asthma according to the Global Initiative for Asthma (GINA) guidelines. Patients will be included at the onset of a (severe) asthma exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Relation of phenotypical characteristics with treatment response | 7 days
  Relation of phenotyipcal characteristics with treatment response defined by 1) the physician - and patient rated global evaluation of treatment effectiveness (GETE) score 2) difference in Asthma Control Questionnaire 5 (ACQ-5) (> 0.5) 3) difference in handheld spirometry values like forced expiratory volume (FEV1 ≥ 10%).

SECONDARY OUTCOMES:
Prediction model for the treatment response of acute asthma exacerbation | 42 days
  Creating a prediction model for the treatment response of acute asthma exacerbation with phenotypical characteristics
Aetiology of the acute asthma exacerbation | 42 days
  Analysing the aetiology of the acute asthma exacerbations
Immune system and microbiome | 42 days
  Analysing the blood and local respiratory parameters; the microbiota composition; lipid metabolomics and volatile compounds composition at baseline and acute asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Gert-Jan Braunstahl, MD, PhD, Principal Investigator — Franciscus Gasthuis & Vlietland; Gerdien Tramper, MD, PhD, Principal Investigator — Franciscus Gasthuis & Vlietland
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided